CLINICAL TRIAL: NCT01519882
Title: A Multi-Centre, Randomized, Double-Blind, Placebo Controlled Study to Evaluate the Effects of Rotigotine on Sleep Efficiency in Patients With Advanced Parkinson's Disease.
Brief Title: Sleep Efficiency Assessed by Polysomnography (PSG Sleep Lab Testing) in Advanced Parkinson's Disease
Acronym: REFRESH-PD
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to major recruitment issues, a decision was made to terminate this trial
Sponsor: UCB Pharma SA (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SP0919; 2011-000056-42 (EudraCT Number)
Record Dates: First submitted 2012-01-24; First posted 2012-01-27 (Estimated); Results first posted 2014-01-28 (Estimated); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Advanced Idiopathic Parkinson's Disease
Keywords: Rotigotine; Neupro; Polysomnography; Sleep efficiency; Advanced Idiopathic Parkinson's Disease; Sleep Disorder
MeSH Terms: conditions — Sleep Wake Disorders | interventions — rotigotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo Transdermal Patches
  Interventions: Other: Placebo
- Rotigotine (Experimental): Rotigotine Transdermal Patches
  Interventions: Other: Rotigotine

INTERVENTIONS:
Other: Placebo — Placebo patches size equivalent to 4, 6 & 8 mg/24 h. Daily application of Placebo patches starting at 4 mg/24 h. Dose will be up-titrated weekly by increments of 2 mg/24 h until optimal or maximal dose is reached. Maximal dose is 16 mg/24 h.
  Optimal or maximal dose will be maintained for 4 Weeks followed by a de-escalation by 2 mg/24 h every other day.
  Arms: Placebo
Other: Rotigotine — Rotigotine patches of 4,6 & 8 mg/24 h. Daily application of Rotigotine patches starting at 4 mg/24 h. Dose will be up-titrated weekly by increments of 2 mg/24 h until optimal or maximal dose is reached. Maximal dose is 16 mg/24 h.
  Optimal or maximal dose will be maintained for 4 weeks followed by a de-escalation by 2 mg/24 h every other day.
  Other Names: Neupro®; (6S)-6-propyl-[2-(2-thienyl)ethyl]amino-5,6,7,8-tetrahydro-1-naphthalenol
  Arms: Rotigotine

SUMMARY:
This is a phase 4 study to evaluate with Polysomnography (PSG) and subjective measures the effect of Rotigotine on sleep efficiency, maintenance, insomnia, nocturnal akinesia and night-time movement in bed, in patients with advanced Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Advanced Parkinson's disease (ie, takes Levodopa (L-DOPA))
* Hoehn and Yahr stage score of 2 to 4
* Subject has sleep-maintenance insomnia

Exclusion Criteria:

* Significant skin disease that would make transdermal drug use inappropriate
* Subject received therapy with controlled-release Levodopa (L-DOPA), entacapone or Stalevo® within 28 days prior to the Baseline Visit or has received therapy with Tolcapone
* Atypical Parkinsonian syndromes
* Previous diagnosis of Narcolepsy, Sleep Apnoea Syndrome, significant Rapid Eye Movement (REM) Sleep Behavior Disorder (RBD), moderate to severe Restless Legs Syndrome (RLS) or Periodic Limb Movement Disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (1):
- 1, Middlesbrough, United Kingdom

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started in March 2012 and was conducted in the United Kingdom. It was terminated due to recruitment issues in January 2013.
Pre-assignment Details: 1 subjects was randomized to Placebo and started and completed the study (from Screening (Week 0) to the Safety Follow-Up Visit (Week 18)).
Groups:
- Placebo: Placebo Transdermal Patches
  Placebo : Placebo patches size equivalent to 4, 6 & 8 mg/24 h. Daily application of Placebo patches starting at 4 mg/24 h. Dose will be up-titrated weekly by increments of 2 mg/24 h until optimal or maximal dose is reached. Maximal dose is 16 mg/24 h.
  Optimal or maximal dose will be maintained for 4 Weeks followed by a de-escalation by 2 mg/24 h every other day.
- Rotigotine: Rotigotine Transdermal Patches
  Rotigotine : Rotigotine patches of 4,6 & 8 mg/24 h. Daily application of Rotigotine patches starting at 4 mg/24 h. Dose will be up-titrated weekly by increments of 2 mg/24 h until optimal or maximal dose is reached. Maximal dose is 16 mg/24 h.
  Optimal or maximal dose will be maintained for 4 weeks followed by a de-escalation by 2 mg/24 h every other day.
Period: Overall Study
Arm/Group | Placebo | Rotigotine
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Rotigotine | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 0 |  | 0
  >=65 years | 1 |  | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (NA) — The mean presented here is the individual age of the only subject included. |  | 67 (NA) — The mean presented here is the individual age of the only subject included.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Sleep Efficiency Index (SEI) to Week 4 of the Maintenance Period
Description: The Sleep Efficiency Index in percent is the ratio of total sleep time (based on Polysomnography recordings) to time in bed (period between "lights off" and "lights on").
Time Frame: From Baseline to Week 4 of the Maintenance Period (up to 11 weeks post-baseline)
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 1 | 0
percentage change | 4.7 (NA) — The mean presented here is the individual percentage change in SEI (from Baseline to Week 4 of the Maintenance Period) of the only subject included. |

2. Secondary Outcome: Change From Baseline in the Parkinson's Disease Sleep Scale Score Version 2 (PDSS2) to Day 1 of the Maintenance Period
Description: The PDSS is a scale to assess sleep and nocturnal disability in Parkinson's Disease during the previous 7 days, and is designed for self-completion by the subject. The updated version (PDSS2) contains 15 questions to be answered using a 5-point Likert scale, where 0 = never, 1 = occasionally, 2 = sometimes, 3 = often, and 4 = very often.
  Thus, PDSS2 score ranges from 0-60, with higher scores indicating worse sleep and higher nocturnal disability. A negative value in Change from Baseline indicates improved sleep and less nocturnal disability.
Time Frame: From Baseline to Day 1 of the Maintenance Period (up to 7 weeks post-baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 1 | 0
units on a scale | 3 (NA) — The mean presented here is the individual change in PDSS2 (from Baseline to Day 1 of the Maintenance Period) of the only subject included. |

3. Secondary Outcome: Change From Baseline in the Parkinson's Disease Sleep Scale Score Version 2 (PDSS2) to Week 4 of the Maintenance Period
Description: The PDSS2 is a scale to assess sleep and nocturnal disability in Parkinson's Disease during the previous 7 days, and is designed for self-completion by the subject. The updated version (PDSS2) contains 15 questions to be answered using a 5-point Likert scale, where 0 = never, 1 = occasionally, 2 = sometimes, 3 = often, and 4 = very often.
  Thus, PDSS2 score ranges from 0-60, with higher scores indicating worse sleep and higher nocturnal disability. A negative value in Change from Baseline indicates improved sleep and less nocturnal disability.
Time Frame: From Baseline to Week 4 of the Maintenance Period (up to 11 weeks post-baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 1 | 0
units on a scale | 6 (NA) — The mean presented here is the individual change in PDSS2 (from Baseline to Week 4 of the Maintenance Period) of the only subject included. |

4. Secondary Outcome: Change From Baseline in the Epworth Sleepiness Score (ESS) to Day 1 of the Maintenance Period
Description: The ESS measures the subject's general level of daytime sleepiness. The 8 items of this scale assess the probability of falling asleep in a variety of situations. Each item is scored by the subject using the following categories:
  0 = would never doze, 1 = slight chance of dozing, 2 = moderate chance of dozing, and 4 = high chance of dozing.
  The ESS score ranges from 0 to 32, with higher values indicating a higher level of daytime sleepiness. A negative value in Change from Baseline indicates a decrease in daytime sleepiness.
Time Frame: From Baseline to Day 1 of the Maintenance Period (up to 7 weeks post-baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 1 | 0
units on a scale | -1 (NA) — The mean presented here is the individual change in ESS (from Baseline to Day 1 of the Maintenance Period) of the only subject included. |

5. Secondary Outcome: Change From Baseline in the Epworth Sleepiness Score (ESS) to Week 4 of the Maintenance Period
Description: as for outcome 4
Time Frame: From Baseline to Week 4 of the Maintenance Period (up to 11 weeks post-baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 1 | 0
units on a scale | 0 (NA) — The mean presented here is the individual change in ESS (from Baseline to Week 4 of the Maintenance Period) of the only subject included. |

6. Secondary Outcome: Change From Baseline in the Sleep Period Time in Non-Rapid Eye Movement (Non-REM) Sleep to Week 4 of the Maintenance Period
Description: Polysomnography (PSG) was performed for the 2 consecutive nights prior to Day 1 and the 2 consecutive nights prior Week 4 of the Maintenance Period.
  Readings from the first night of the PSG will not be used for analysis as this is considered an adaptation night.
  The subject was not allowed to sleep during the daytime on the day of a PSG reading. The PSG was recorded for a minimum of 6 h and a maximum of 8 h.
  The sleep period time in stage 3 non-REM was derived from the hypnogram, based on Electroencephalogram (EEG), Electro-myogram (EMG), Electro-oculogram (EOG) and Electrocardiogram (ECG). Change from Baseline is calculated by:
  (Stage 3 non-REM time (in minutes) at Baseline)- (Stage 3 non-REM time (in minutes) at Week 4 of the MP).
Time Frame: From Baseline to Week 4 of the Maintenance Period (up to 11 weeks post-baseline)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 1 | 0
minutes | 22 (NA) — The mean presented here is the individual change in sleep Period time in Non-REM sleep (from Baseline to Week 4 of the Maintenance Period) of the only subject included. |

7. Secondary Outcome: Change From Baseline in the Nocturnal Akinesia, Dystonia, and Cramps Score (NADCS) to Day 1 of the Maintenance Period
Description: The NADCS assesses nocturnal akinesia, dystonia, and cramps using an ordinal severity scale. While a score of 0 = normal and 4 = maximal severity, subjects can also rate their symptoms with values of 0.5, 1.5, 2.5, and 3.5. The nocturnal akinesia score was used to evaluate motor performance while the dystonia and cramps score was used to evaluate pain. A negative value in Change from Baseline indicates an improvement.
Time Frame: From Baseline to Day 1 of the Maintenance Period (up to 7 weeks post-baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 1 | 0
units on a scale | -0.5 (NA) — The mean presented here is the individual change in NADCS (from Baseline to Day 1 of the Maintenance Period) of the only subject included. |

8. Secondary Outcome: Change From Baseline in the Nocturnal Akinesia, Dystonia and Cramps Score (NADCS) to Week 4 of the Maintenance Period
Description: as for outcome 7
Time Frame: From Baseline to Week 4 of the Maintenance Period (up to 11 weeks post-baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 1 | 0
units on a scale | -0.5 (NA) — The mean presented here is the individual change in NADCS (from Baseline to Week 4 of the Maintenance Period) of the only subject included. |

9. Secondary Outcome: Change From Baseline in the Total Wake Time After Sleep Onset (WASO) to Week 4 of the Maintenance Period
Description: Polysomnography (PSG) was performed for the 2 consecutive nights prior to Day 1 and the 2 consecutive nights prior Week 4 of the Maintenance Period.
  Readings from the first night of the PSG will not be used for analysis as this is considered an adaptation night.
  The subject was not allowed to sleep during the daytime on the day of a PSG reading. The PSG was recorded for a minimum of 6 h and a maximum of 8 h.
  Sleep stages and time spent in each sleep stage were determined from EEG readings. WASO was calculated by:
  (Time in bed (Period between "lights off" and "lights on"))-(Sleep time).
Time Frame: From Baseline to Week 4 of the Maintenance Period (up to 11 weeks post-baseline)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 1 | 0
minutes | 20 (NA) — The mean presented here is the individual change in total Wake Time After Sleep Onset (from Baseline to Week 4 of the Maintenance Period) of the only subject included. |

10. Secondary Outcome: Change From Baseline in the Total Number of Turnings in Bed to Week 4 of the Maintenance Period
Description: Polysomnography (PSG) was performed for the 2 consecutive nights prior to Day 1 and the 2 consecutive nights prior Week 4 of the Maintenance Period.
  Readings from the first night of the PSG will not be used for analysis as this is considered an adaptation night.
  The subject was not allowed to sleep during the daytime on the day of a PSG reading. The PSG was recorded for a minimum of 6 h and a maximum of 8 h.
  The number of turnings in bed was determined via a postural sensor placed on the subject's chest.
Time Frame: From Baseline to Week 4 of the Maintenance Period (up to 11 weeks post-baseline)
Measure: Number; unit: Number of turnings in bed
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 1 | 0
Number of turnings in bed | 0 |

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from Baseline to the Safety Follow-Up Visit at Week 18.
Arm/Group | Placebo | Rotigotine
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=1) | Rotigotine (N=0)
Constipation (Gastrointestinal disorders) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Tension Headache (Nervous system disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Despite many attempts by study sites to recruit subjects, only 1 subject was randomized by Oct 2012. The decision to terminate the study was taken in Nov 2012. The subject completed in Jan 2013.

No planned efficacy/safety analyses were performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days